CLINICAL TRIAL: NCT02443233
Title: Evaluation of Paternal, Maternal and Obstetric Factors Leading to the Hepatitis B Immunization Failure in Hong Kong
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 13-270
Record Dates: First submitted 2015-04-28; First posted 2015-05-13 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B Infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Maternal hepatitis B carrier
- Paternal hepatitis B carrier

SUMMARY:
Globally, hepatitis B virus (HBV) infection is the most common form of chronic hepatitis. There are still a lot of uncertainties on how infants acquired HBV leading to the development of chronic HBV infection despite active and passive immunoprophylaxis. The investigators would like to carry out a prospective study to answer the following questions:

1. the paternal, maternal and obstetric factors leading to immunoprophylaxis failure
2. the prevalence of immunoprophylaxis failure in Hong Kong

ELIGIBILITY:
Inclusion Criteria:

* All women age ≥ 18 years
* Maternal or paternal hepatitis B carrier

Exclusion Criteria:

* Couples will be excluded if female partners of paternal hepatitis B carrier were occult carrier
* Plan to deliver in other units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Maternal and paternal hepatitis B carrier
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The effect of high maternal viral load on immunoprophylaxis failure, using 10^6 copies/ml as cut-off | Infants' blood for HbsAg at 9-12 months old

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wang Cheung, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China